CLINICAL TRIAL: NCT04828967
Title: The Effect of Adjuvant Hypnosis Added to Conventional Therapy on Nausea and Vomiting in Hyperemesis Gravidarum: A Prospective Randomized Study
Brief Title: Use of Hypnosis in Hyperemesis Gravidarum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyda Efsun Ozgunay, Assoc Prof, Turkiye Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 66519339-900-01/2015/02-04
Record Dates: First submitted 2021-03-27; First posted 2021-04-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Nausea; Vomiting; Hyperemesis Gravidarum
Keywords: hyperemesis gravidarum; hypnosis; nausea
MeSH Terms: conditions — Nausea; Vomiting; Hyperemesis Gravidarum | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental): Hypnosis is added to the conventional group.
  Interventions: Other: Hypnosis
- conventional group (No Intervention): only conventional group

INTERVENTIONS:
Other: Hypnosis — Hypnosis is added to the conventional group
  Other Names: Conventionel
  Arms: Hypnosis group

SUMMARY:
Aim: It has been aimed in this study to investigate the effects of hypnosis used to augment the conventional therapy on nausea, vomiting, rescue drug consumption and hospital stay in cases of Hyperemesis Gravidarum (HG).

Methods: This prospective randomised study was carried out with 41 inpatients diagnosed with HG. The patients were grouped as GH (n=18) given hypnosis and GC (n=23) not given hypnosis with the conventional therapy. Group H were hypnotized during two sessions and taught auto-hypnosis. Data on the patient demographics, VAS scores for severity of nausea, the numbers of vomiting per day, additional medications used and the days of hospital stay were recorded.

DETAILED DESCRIPTION:
This prospective, randomised and single blind study, with the physician follow up the patients for nausea and vomiting not informed on the grouping of the patients, was carried out at a single center between January 2017 and January 2018. The study protocol was approved by the local Ethics Committee was conducted in accordance with the principles of the Declaration of Helsinki Written informed consent was obtained from the patients.

Pregnant patients above the age of 18 years, admitted to the hospital with HG diagnosis were included in the study. HG was diagnosed on the basis of having at least one of the symptoms of ketonuria, weight loss in excess of 5% of the body weight and serious vomiting more than twice per day. Patients with known psychiatric disorders, organic diseases causing nausea and vomiting, HG diagnosis in previous pregnancy and experience in hypnosis, meditation and mindfullness, and those who were multiparous or could not be cooperative with the treatment team were excluded from the study.

The patients were randomly assigned by means of picking closed envolopes to the Group H (GH) to receive hypnosis with conventional therapy and the Group C (GC) only to receive conventional therapy. Data on patient demographics, severity of nausea, numbers of vomiting per day, serum glucose, AST and ALT levels were recorded. Nausea and vomiting severity were evaluated 4 times per day using the Visual Analog Scale (VAS 0-10; with 0=no nausea and10=extreme nausea).

Conventional Ttreatment The treatment in HG is targeted to minimise the symptoms in order to reduce the adverse outcomes for the mother and the foetus. In our study, the conventional treatment was organized according to symptom severity, the clinical findings and the response given to the treatment. The basic protocol for the first 24 hours included intravenous hydration for 6 hours with NaCl (0.9 % x1000 cc) supplemented with KCL, the B1 and B6 vitamins. Oral feeding was restricted and the second step treatment choice comprising H1 receptor blocker dimenhydrinate (4 X 50 mg/day, po) was routinely used in all patients. When the VAS score was ≥4, the serotonin antagonist ondansetron (4mg, i.v.) was added to the treatment as the rescue medication. The daily nausea, numbers of vomiting were queried on a daily basis. The patients with vomiting incidence below 2 per day, tolerating oral nutrition and with urine cleared of ketonuria met the conditions of discharge. The duration of hospital stay and treatment procedures were followed and recorded.

Hypnosis design Two sessions of hypnosis were carried out in addition to the conventional treatment on the first and second days of admission; and the paitents were instructed autohypnosis after the second session. This was repeated on the third day with the patients who could not satisfactorily acquire the technique and those who failed to succeed were excluded from the study. The GH included patients who carried out autohypnosis minimally 4 times per day.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients above the age of 18 years, admitted to the hospital with HG diagnosis were included in the study. HG was diagnosed on the basis of having at least one of the symptoms of ketonuria, weight loss in excess of 5% of the body weight and serious vomiting more than twice per day.

Exclusion Criteria:

* Patients with known psychiatric disorders, organic diseases causing nausea and vomiting, HG diagnosis in previous pregnancy and experience in hypnosis, meditation and mindfulness, and those who were multiparous or could not be cooperative with the treatment team were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
The Effect of Adjuvant Hypnosis on Nausea and Vomiting in Hyperemesis Gravidarum | baseline + 12 months
  Data on severity of nausea, numbers of vomiting per day were recorded. Deducting the score at discharge from the score at arrival indicated the decrease in the VAS score during treatment. Nausea and vomiting severity were evaluated 4 times per day using the Visual Analog Scale (VAS 0-10; with 0=no nausea and10=extreme nausea).

SECONDARY OUTCOMES:
The effect of hypnosis on hospital stay | baseline + 12 months
  To obtain data on the severity of nausea, the daily number of vomiting. To determine the difference between VAS value during discharge and VAS ariviing hospitalization. Nausea and vomiting severity were evaluated 4 times a day using theVisual Analogue Scale (VAS 0-10; 0 = no nausea and 10 = excessive nausea).

CONTACTS AND LOCATIONS:
Overall Officials: Seyda E Ozgunay, Principal Investigator — Bursa Yuksek ihtisas research and training hospital; Burcu Cakmak, Principal Investigator — Bursa Yuksek ihtisas research and training hospital
Locations (1):
- Bursa yuksek ihtisas eğitim araştırma hastanesi, Bursa, Yildirim/Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Philip B. Hyperemesis gravidarum: literature review. WMJ. 2003;102(3):46-51. PMID 12822290
- [Result] Wegrzyniak LJ, Repke JT, Ural SH. Treatment of hyperemesis gravidarum. Rev Obstet Gynecol. 2012;5(2):78-84. PMID 22866186
- [Result] Tan PC, Omar SZ. Contemporary approaches to hyperemesis during pregnancy. Curr Opin Obstet Gynecol. 2011 Apr;23(2):87-93. doi: 10.1097/GCO.0b013e328342d208. PMID 21297474
- [Result] Ergin M, Cendek BD, Neselioglu S, Avsar AF, Erel O. Dynamic thiol-disulfide homeostasis in hyperemesis gravidarum. J Perinatol. 2015 Oct;35(10):788-92. doi: 10.1038/jp.2015.81. Epub 2015 Jul 9. PMID 26156064
- [Result] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Result] Werner A, Uldbjerg N, Zachariae R, Nohr EA. Effect of self-hypnosis on duration of labor and maternal and neonatal outcomes: a randomized controlled trial. Acta Obstet Gynecol Scand. 2013 Jul;92(7):816-23. doi: 10.1111/aogs.12141. Epub 2013 Apr 22. PMID 23550694
- [Result] Longo F, Mansueto G, Lapadula V, Stumbo L, Del Bene G, Adua D, De Filippis L, Bonizzoni E, Quadrini S. Combination of aprepitant, palonosetron and dexamethasone as antiemetic prophylaxis in lung cancer patients receiving multiple cycles of cisplatin-based chemotherapy. Int J Clin Pract. 2012 Aug;66(8):753-757. doi: 10.1111/j.1742-1241.2012.02969.x. Epub 2012 Jul 2. PMID 22805267
- [Result] Emami-Sahebi A, Elyasi F, Yazdani-Charati J, Shahhosseini Z. Psychological interventions for nausea and vomiting of pregnancy: A systematic review. Taiwan J Obstet Gynecol. 2018 Oct;57(5):644-649. doi: 10.1016/j.tjog.2018.08.005. PMID 30342643